CLINICAL TRIAL: NCT06516328
Title: AGE/sRAGE and IL-17 Levels in Type 2 Diabetic Periodontitis Patients
Brief Title: AGE/sRAGE Ratio in Diabetic Periodontitis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yagmur Deniz YILDIRIM, Asistant Proffessor, Hacettepe University
Other Study IDs: GO23/63
Record Dates: First submitted 2024-07-14; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis, Diabetes Mellitus Type 2
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy (H): Periodontally and systemically healthy individuals
  Interventions: Other: Observational
- Periodontitis (P): Patients with periodontitis without diabetes
  Interventions: Other: Observational
- Diabetic Periodontitis (DP) group: Periodontitis patients with diabetes under control (Glycosylated hemoglobin (HbA1c) value ≤ 6.5% and fasting blood sugar levels <200 mg/dl.)
  Interventions: Other: Observational
- Poorly controlled Diabetic Periodontitis group (PDP): Periodontitis patients with uncontrolled diabetes HbA1c value > 6.5% and fasting blood sugar levels > 200 mg/dl.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — GCF and saliva samples obtained.

SUMMARY:
The goal of this observational study is to learn about some molecules in the disease mechanism of type 2 diabetes and periodontitis. There are end products inside the body called AGEs and their receptors binding to them especially (sRAGE, RAGE) in people with diabetes in hyperglycemic state.These molecules are important also in periodontitis (the disease of teeth that may end with exfoliation of the tooth). Diabetes and periodontitis enhance each other's disease-causing effects. Both is chronic inflammatory diseases and IL-17 is another molecule having role in this process.

Totally 64 men and women aged between 27-60 included in the study. Study groups were : 1.participants with healthy teeth and no diabetes, 2. participants with periodontitis without diabetes, 3.participants with periodontitis and controlled diabetes, 4.participants with periodontitis and uncontrolled diabetes (6.5% and fasting blood sugar levels <200 mg/dl). Researchers got saliva and gingival crevicular fluid (GCF) samples from diseased teeth and examined AGE, sRAGE, IL-17 levels. GCF is a fluid around the crevice of the theeth with different characteristics from saliva.

As a result AGE/sRAGE ratio and IL-17 levels of diseased groups were higher than healthy group, while sRAGE levels were significantly lower in GCF samples. Researchers concluded that GCF and saliva AGE/sRAGE ratio may represent as a biomarker in periodontitis patients with uncontrolled diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Having interdental attachment loss in at least two non-adjacent teeth, or with >3 mm of attachment loss in the buccal or palatal/lingual region with >3 mm probing depth in at least two teeth for periodontitis groups.
* Having minimum 5mm or more pocket depth in at least 6 periodontal pockets.
* HbA1c value ≤ 6.5% and fasting blood sugar levels <200 mg/dl for the controlled diabetes group.
* HbA1c value > 6.5% and fasting blood sugar levels > 200 mg/dl for uncontrolled diabetes group.

Exclusion Criteria:

* having periodontal treatment in the last six months;
* participants with smoking habit or history; and
* usage of medicine that may affect study results (mouthwash, antibiotics, corticosteroid, statins etc.) three months before collecting dental plaque and GCF samples.
* Lactating or pregnant patients
* Patients with systemic diseases other than type 2 diabetes.

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of participants who applied to Hacettepe University Department of Periodontology and Hacettepe University Department of Endocrinology and Metabolism. Patients who agreed to participate in the study gave their written informed consent were included.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
AGEs/RAGE ratio, IL-17 level in GCF and saliva | 3 to 6 months
  AGEs to RAGE ratio comparison between study groups
AGEs/RAGE ratio, IL-17 level in GCF and saliva | 3 to 6 months
  IL-17 level comparison between study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)